CLINICAL TRIAL: NCT02952508
Title: An Open-Label, Multicenter, Phase 2 Study of Iopofosine I 131 (CLR 131) in Patients With Relapsed or Refractory (R/R) Select B-Cell Malignancies (CLOVER-1) and Expansion Cohort in Patients With Waldenstrom Macroglobulinemia (CLOVER-WaM)
Brief Title: Study of Iopofosine I 131 (CLR 131) in Select B-Cell Malignancies (CLOVER-1) and Pivotal Expansion in Waldenstrom Macroglobulinemia
Acronym: CLOVER-WaM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCL-16-001
Record Dates: First submitted 2016-10-28; First posted 2016-11-02 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2024-09

CONDITIONS: Waldenstrom Macroglobulinemia; Multiple Myeloma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma; Central Nervous System Lymphoma
Keywords: Waldenstrom Macroglobulinemia; Non-Hodgkin Lymphoma; NHL; Relapsed; Refractory; Novel class; Pivotal; Phase 3; Hematologic disease; Neoplasm; Plasma cell neoplasms; Paraproteinemias; Lymphoma; Immunoproliferative disorder; Blood protein disorders; Lymphoproliferative disorders; Antineoplastic agents
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Recurrence; Hematologic Diseases; Neoplasms; Neoplasms, Plasma Cell; Paraproteinemias; Lymphoma; Immunoproliferative Disorders; Blood Protein Disorders; Lymphoproliferative Disorders | interventions — CLR1404

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Iopofosine I 131, intravenous administration WM (Experimental): Iopofosine I 131 in Waldenstroms Macroglobulinemia
  Interventions: Drug: Iopofosine I 131 single dose; Drug: Iopofosine I 131 multiple dose; Drug: Iopofosine I 131 fractionated dose
- Iopofosine I 131, intravenous administration MM (Experimental): Iopofosine I 131 in Multiple Myeloma
  Interventions: Drug: Iopofosine I 131 single dose; Drug: Iopofosine I 131 multiple dose; Drug: Iopofosine I 131 fractionated dose
- Iopofosine I 131, intravenous administration CNS Lymphoma (Experimental): Iopofosine I 131 in Central Nervous System Lymphoma
  Interventions: Drug: Iopofosine I 131 fractionated dose
- Iopofosine I 131 intravenous administration NHL [CLOSED] (Experimental): Iopofosine I 131 in Chronic Lymphocytic Leukemia / Small Lymphocytic Lymphoma, Mantle Cell Lymphoma, Marginal Zone Lymphoma, and Diffuse Large B-Cell Lymphoma
  Interventions: Drug: Iopofosine I 131 single dose; Drug: Iopofosine I 131 multiple dose; Drug: Iopofosine I 131 fractionated dose

INTERVENTIONS:
Drug: Iopofosine I 131 single dose — Radiopharmaceutical
  Other Names: I-131-CLR1404; CLR 131
  Arms: Iopofosine I 131 intravenous administration NHL [CLOSED]; Iopofosine I 131, intravenous administration MM; Iopofosine I 131, intravenous administration WM
Drug: Iopofosine I 131 multiple dose — Radiopharmaceutical
  Other Names: I-131-CLR1404; CLR 131
  Arms: Iopofosine I 131 intravenous administration NHL [CLOSED]; Iopofosine I 131, intravenous administration MM; Iopofosine I 131, intravenous administration WM
Drug: Iopofosine I 131 fractionated dose — Radiopharmaceutical
  Other Names: I-131-CLR1404; CLR 131

SUMMARY:
Part A of this study evaluates iopofosine I 131 (CLR 131) in patients with select B-cell malignancies (multiple myeloma( MM), indolent chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), lymphoplasmacytic lymphoma (LPL)/Waldenstrom Macroglobulinemia (WM), marginal zone lymphoma (MZL), mantle cell lymphoma (MCL), diffuse large B-cell lymphoma (DLBCL), and central nervous system lymphoma (CNSL) who have been previously treated with standard therapy for their underlying malignancy. Part B (CLOVER-WaM) is a pivotal efficacy study evaluating IV administration of iopofosine I 131 in patients with WM that have received at least two prior lines of therapy.

DETAILED DESCRIPTION:
B-cell malignancies represent a diverse collection of diseases and, taken together, make up the majority of hematologic malignancies. B-cell lymphomas represent the largest percentage of these neoplasms, and the relapsed and/or refractory B-cell lymphomas have proven very difficult to treat. Patients that have failed prior therapy, including WM patients, represent a very challenging patient population with significantly reduced life-expectancy.

Iopofosine I 131 is a targeted radiotherapeutic that exploits the selective uptake and retention of Cellectar's proprietary phospholipid ethers (PLEs) by malignant cells. Cellectar Biosciences' novel cancer-targeted small-molecule compound is radiolabeled with the radioisotope iodine-131 (I-131) which has previously been used approved for use in select tumors. Iopofosine I 131 has been evaluated in over 80 xenograft and spontaneous (transgenic) tumor models where it was demonstrated to be effective in eliminating tumors.

Based on the critical unmet medical need for effective agents with novel mechanisms of action in B-cell malignancies, Cellectar Biosciences has chosen to expand this ongoing study to assess iopofosine I 131 in a pivotal expansion cohort in Waldenstrom's Macroglobulinemia patients that have received at least two prior lines of therapy.

ELIGIBILITY:
[CLOVER-1] Inclusion Criteria: All Patients

* Histologically or cytologically confirmed MM; Patients with primary or secondary CNSL may be enrolled.
* ECOG performance status of 0 to 2
* 18 years of age or older
* Life expectancy of at least 6 months
* Platelets ≥ 75,000/µL (if full-dose anticoagulation therapy is used, platelets ≥ 100,000/µL are required)
* WBC count ≥ 3000/µL
* Absolute neutrophil count ≥ 1500/µL
* Hemoglobin ≥ 9 g/dL (last transfusion, if any, must be at least 1 week prior to study registration, and no transfusions are allowed between registration and dosing)
* Estimated glomerular filtration rate ≥ 30 mL/min/1.73 m2
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN)
* Bilirubin < 1.5 × ULN
* International normalized ratio (INR) < 2.5
* If patient is on full-dose anticoagulation therapy, the anticoagulation therapy must be reversible and reversal of the anticoagulation therapy must not be life-threatening, as judged by the Investigator
* Patients who have undergone stem cell transplant must be at least 100 days from transplant

Patients with Multiple Myeloma

* At least 5 prior regimens, which must include at least 1 approved proteasome inhibitor (bortezomib, carfilzomib, or ixazomib), at least 1 approved immunomodulatory agent (thalidomide, lenalidomide, or pomalidomide), and at least 1 approved monoclonal antibody (e.g., daratumumab or elotuzumab) with or without maintenance therapy, unless patients are intolerable to such agents or ineligible to receive such agents.
* At least triple-class refractory (refractory to a proteasome inhibitor, immunomodulatory agent, and a monoclonal antibody)
* Progressive disease defined by any of the following:

  * 25% increase in serum M-protein from the lowest response value during (or after) last therapy and/or absolute increase in serum M-protein of ≥ 0.5 g/dL
  * 25% increase in urine M-protein from the lowest response value during (or after) last therapy and/or absolute increase in urine M-protein of ≥ 200 mg/24 h
  * 25% increase in bone marrow plasma cell percentage from the lowest response value during (or after) last therapy. Absolute bone marrow plasma cell percentage must be ≥ 10% unless prior CR when absolute bone marrow plasma cell percentage must be ≥ 5%.
  * 25% increase in serum FLC level from the lowest response value during (or after) last therapy; the absolute increase must be > 10 mg/dL
  * New onset hypercalcemia > 11.5 mg/dL
  * Failure to obtain a partial response or better to current treatment, or cannot further improve their response to current treatment
  * Appearance of new extramedullary disease
* Measurable disease defined by any of the following:

  * Serum M-protein > 0.5 g/dL
  * Urine M-protein > 200 mg/24 h
  * Serum FLC assay: Involved FLC level ≥ 10 mg/dL provided serum FLC ratio is abnormal.

[CLOSED] Patients with Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma, Lymphoplasmacytic Lymphoma/Waldenstom Macroglobulinemia, or Marginal Zone Lymphoma

* Prior treatment with at least 2 prior regimens, which may include chemotherapy, an approved anti-CD20 antibody with or without maintenance therapy, and an approved targeted agent, unless patients are ineligible to receive such agents
* Patients with Helicobacter pylori+ mucosa-associated lymphoid tissue lymphoma must have received 1 prior antibiotic regimen for H pylori
* At least 1 measurable nodal lesion with longest diameter > 15 mm or 1 measurable extranodal lesion (eg, hepatic nodule) with longest diameter > 10 mm. Additional parameters (e.g., measurable IgM for patients with Lymphoplasmacytic Lymphoma) may be allowed if they meet current NCCN guidelines for symptomatic disease. Patients with uptake by FDG-PET scan may be allowed with prior approval of Sponsor.

[CLOSED] Patients with Mantle Cell Lymphoma

* Prior treatment with at least 1 prior regimen
* At least 1 measurable nodal lesion with longest diameter > 15 mm or 1 measurable extranodal lesion (eg, hepatic nodule) with longest diameter > 10 mm. Patients with uptake by FDG-PET scan may be allowed with prior approval of Sponsor.

[CLOSED] Patients with Diffuse Large B-Cell Lymphoma

* Relapsed or refractory to combination chemotherapy for DLBCL that contains rituximab and an anthracycline; or is intolerable to such agents. Relapsed disease is defined as either recurrence of disease after a CR or PD after achieving a partial response (PR) or SD. Refractory disease is defined as failure to achieve at least SD with any 1 line of therapy or with PD ≤ 3 months of the most recent chemotherapy regimen.
* At least 1 measurable nodal lesion with longest diameter > 15 mm or 1 measurable extranodal lesion (eg, hepatic nodule) with longest diameter > 10 mm. Patients with uptake by FDG-PET scan may be allowed with prior approval of Sponsor.

Patients with CNS Lymphoma

* Must have biopsy-proven disease and must have received at least one prior intervention for their disease.
* Must be at least two weeks from CNS biopsy before administration of iopofosine I 131.
* Must have at least one lesion with enhancement on brain imaging.
* Stable (or decreasing) dose of corticosteroids or anti-convulsant medication for at least 7 days prior to dosing

[CLOVER-1] Exclusion Criteria:

* Ongoing Grade 2 or greater toxicities due to previous therapies. Stable, tolerable Grade 2 AEs (eg, neuropathy) may be allowed.
* Prior external-beam RT resulting in greater than 20% of total bone marrow receiving greater than 20 Gy.
* Prior total body or hemi-body irradiation. Patients who have received prior low-dose total body or hemi-body irradiation may be allowed on a case-by-case basis after discussion with Sponsor (considerations may include factors such as time since irradiation, total lifetime accumulated dose, etc.)
* Extradural tumor in contact with the spinal cord or tumor located where swelling in response to therapy may impinge upon the spinal cord
* For patients with CLL/SLL, LPL, or MZL, transformation to a more aggressive form of NHL
* Ongoing chronic immunosuppressive therapy
* Clinically significant bleeding event within prior 6 months
* Ongoing anti-platelet therapy (except low-dose aspirin [eg, 81 mg daily] for cardioprotection)
* Anti-cancer therapy within two weeks of initial iopofosine I 131 infusion. Low dose dexamethasone for symptom management is allowed
* Radiation therapy, chemotherapy, immunotherapy, or investigational therapy within 2 weeks of eligibility-defining bone marrow biopsy.
* For patients with primary or secondary CNSL, active bleeding in the tumor bed and/or uncontrolled seizure activity

[CLOVER-WaM] Inclusion Criteria

* Histologically or cytologically confirmed WM. Patients with a diagnosis of LPL may be enrolled with prior Sponsor approval.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2 (Appendix C)
* Patient is 18 years of age or older
* Life expectancy of at least 6 months
* Received at least two prior lines of therapy for WM
* Measurable IgM (above upper limit of normal) OR at least one measurable nodal lesion with longest diameter > 15 mm or one measurable extranodal lesion (e.g., hepatic nodule) with longest diameter > 10 mm

[CLOVER-WaM] Exclusion Criteria

* Ongoing Grade 2 or greater toxicities due to previous therapies, excluding alopecia.
* Prior external-beam RT resulting in greater than 20% of total bone marrow receiving greater than 20 Gy.
* Prior total body or hemi-body irradiation. Patients who have received prior low-dose total body or hemi-body irradiation may be allowed on a case-by-case basis after discussion with Sponsor (considerations may include factors such as time since irradiation, total lifetime accumulated dose, etc.)
* Patients with second malignancies in addition to WM, if the second malignancy has required therapy in the last 2 years or is not in remission; exceptions to this criterion include successfully treated non-metastatic basal cell or squamous cell skin carcinoma, or prostate cancer that does not require therapy
* Anti-cancer therapy within two weeks of initial iopofosine I 131 infusion.
* Need for acute treatment of WM (e.g., those with hyperviscosity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Part A [CLOVER-1] Clinical benefit rate | 84 days
  Response assessment per International Uniform Response Criteria for Multiple Myeloma; Lugano Criteria for lymphoma; International Workshop on Chronic Lymphocytic Leukemia for CLL; VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment; or 2005 Response Criteria for CNS Lymphoma
Part B [CLOVER-WaM] Major Response Rate | 12 months
  Response assessment per criteria modified from VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment

SECONDARY OUTCOMES:
Part A [CLOVER-1] Overall Response Rate | 135 days
  Response assessment per International Uniform Response Criteria for Multiple Myeloma; Lugano Criteria for lymphoma; International Workshop on Chronic Lymphocytic Leukemia for CLL; VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment; or 2005 Response Criteria for CNS Lymphoma
Part A [CLOVER-1] Progression Free Survival | 135 days
  Response assessment per International Uniform Response Criteria for Multiple Myeloma; Lugano Criteria for lymphoma; International Workshop on Chronic Lymphocytic Leukemia for CLL; VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment; or 2005 Response Criteria for CNS Lymphoma
Part A [CLOVER-1] Time to Next Treatment | 3 years
  Response assessment per International Uniform Response Criteria for Multiple Myeloma; Lugano Criteria for lymphoma; International Workshop on Chronic Lymphocytic Leukemia for CLL; VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment; or 2005 Response Criteria for CNS Lymphoma
Part A [CLOVER-1] Overall Survival | 135 days
  Response assessment per International Uniform Response Criteria for Multiple Myeloma; Lugano Criteria for lymphoma; International Workshop on Chronic Lymphocytic Leukemia for CLL; VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment; or 2005 Response Criteria for CNS Lymphoma
Part A [CLOVER-1] Duration of Response | 135 days
  Response assessment per International Uniform Response Criteria for Multiple Myeloma; Lugano Criteria for lymphoma; International Workshop on Chronic Lymphocytic Leukemia for CLL; VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment; or 2005 Response Criteria for CNS Lymphoma
Part B [CLOVER-WaM] Overall Response Rate | 135 days
  Response assessment per criteria modified from VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment
Part B [CLOVER-WaM] Treatment Free Survival | 135 days
  Response assessment per criteria modified from VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment
Part B [CLOVER-WaM] Duration of Response | 135 days
  Response assessment per criteria modified from VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment
Part B [CLOVER-WaM] Clinical Benefit Rate | 135 days
  Response assessment per criteria modified from VIth Waldenstrom's Macroglobulinemia Criteria for Response Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jarrod Longcor, Study Director — Cellectar Biosciences
Locations (50):
- United States (28):
  - Cellectar Biosciences site, Los Angeles, California
  - Cellectar Biosciences site, Redlands, California
  - Cellectar Biosciences site, Washington D.C., District of Columbia
  - Cellectar Biosciences site, Jacksonville, Florida
  - Cellectar Biosciences site, Miami, Florida
  - Cellectar Biosciences site, Tampa, Florida
  - Cellectar Biosciences, Atlanta, Georgia
  - Cellectar Biosciences site, Maywood, Illinois
  - Cellectar Biosciences site, Warrenville, Illinois
  - Cellectar Biosciences site, Westwood, Kansas
  - Cellectar Biosciences site, New Orleans, Louisiana
  - Cellectar Biosciences site, Baltimore, Maryland
  - Cellectar Biosciences, Bethesda, Maryland
  - Cellectar Biosciences site, Boston, Massachusetts
  - Cellectar Biosciences, North Bergen, New Jersey
  - Cellectar Biosciences site, Buffalo, New York
  - Cellectar Biosciences site, New York, New York
  - Cellectar Biosciences site, Rochester, New York
  - Cellectar Biosciences site, Durham, North Carolina
  - Cellectar Biosciences, Canton, Ohio
  - Cellectar Biosciences site, Cincinnati, Ohio
  - Cellectar Biosciences Site, Charleston, South Carolina
  - Cellectar Biosciences, Greenville, South Carolina
  - Cellectar Biosciences site, Knoxville, Tennessee
  - Cellectar Biosciences site, Dallas, Texas
  - Cellectar Biosciences site, Houston, Texas
  - Cellectar Biosciences site, Seattle, Washington
  - Cellectar Biosciences site, Madison, Wisconsin
- Australia (2):
  - Cellectar Biosciences site, Concord, New South Wales
  - Cellectar Biosciences, Adelaide, South Australia
- Brazil (4):
  - Cellectar Biosciences, Salvador, Estado de Bahia
  - Cellectar Biosciences, Curitiba, Paraná
  - Cellectar Biosciences, Porto Alegre, RioGrande Do Sul
  - Cellectar Biosciences, Blumenau, Santa Catarina
- Cellectar Biosciences Site, Hradec Králové, Czechia
- Cellectar Biosciences, Helsinki, Finland
- France (2):
  - Cellectar Biosciences, Pessac
  - Cellectar Biosciences, Poitiers
- Greece (2):
  - Cellectar Biosciences site, Athens
  - Cellectar Biosciences Site, Rio
- Cellectar Biosciences Site, Jerusalem, Israel
- Spain (5):
  - Cellectar Biosciences, Barcelona
  - Cellectar Biosciences site, Barcelona
  - Cellectar Biosciences, Madrid
  - Cellectar Biosciences, Salamanca
  - Cellectar Biosciences site, Zaragoza
- Turkey (Türkiye) (3):
  - Cellectar Biosciences, Ankara
  - Cellectar Biosciences, Bornova
  - Cellectar Biosciences, Istanbul
- Cellectar Biosciences site, London, United Kingdom